CLINICAL TRIAL: NCT00368433
Title: Hypersensitivity in Tourette Syndrome: An Evaluation of Perceived Intensity Versus Threshold
Brief Title: Hypersensitivity in Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060232; 06-N-0232
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-24

CONDITIONS: Tourette's Syndrome
Keywords: Sensory Processing; Electromyogram; Tic Disorder; Tourette Syndrome; Tourette's Syndrome; Healthy Volunteer; HV
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

SUMMARY:
This study will investigate how the sensitivity to touch and smell in patients with Tourette syndrome (TS) may differ from that of people without TS. TS is a neurological disorder that causes people to have uncontrolled movements called "tics." A tic can also be vocal, like a cough or bark or string of bad words. The tic is preceded by a "premonitory urge" that may feel like an itch or pressure that builds until the tic occurs. To some patients, the tic feels like a response to an involuntary sensation. In patients with TS, sensory information may be processed differently than it is in people without TS. This study will compare how strong a sensation feels in TS patients and healthy volunteers. It will also look for muscle activity that may be responsible for the feelings in the area of the tic.

Healthy normal volunteers and people with Tourette syndrome, 18 to 65 years of age, may be eligible for this study. Candidates are screened with a medical history and brief physical and neurological examinations. TS patients complete a questionnaire about their tics and are interviewed by a psychiatrist. Women who can become pregnant will have a urine pregnancy test prior to any other procedures. Pregnant women cannot participate.

All participants undergo sensory testing for touch and smell. They are asked to distinguish between a scented and scentless object and rate how strongly they feel the scent. Later, with their eyes closed, they are asked to tell whether or not they are being touched, and to rate how intensely they felt the touch.

In addition to the sensory testing, TS patients, but not normal volunteers, undergo electromyography (EMG), a test that measures the electrical activity of muscles. For surface EMG, small metal disks called electrodes are filled with a conductive gel and taped to the skin. Wire EMG involves inserting a wire into a muscle using a needle. All patients have surface EMG and those who consent to it will also have wire EMG.

DETAILED DESCRIPTION:
OBJECTIVE:

This study will explore sensory phenomena associated with Tourette syndrome (TS). The first part will evaluate threshold levels versus perceived intensity of tactile and olfactory stimuli in areas reported to be hypersensitive in TS patients. The second part will use electromyography (EMG) to seek correlation between muscle activity and the perceived intensity of "urge" in focal areas of premonitory sensations.

STUDY POPULATION:

Twenty-six patients and 22 control subjects will be studied. Subjects can be of any race, gender, handedness, or age from 18 to 65 years.

DESIGN:

To determine olfactory and tactile threshold, n-butanol and Von Frey hairs will be presented in forced-choice modified method of limits paradigms. Perceived intensity will be examined using a generalized labeled magnitude scale (gLMS), whose word values are placed on a ruler for numerical reporting. Randomly arranged series of 7 stimuli for olfaction and touch will be presented in 4 sets, and subjects will report a number on the gLMS that corresponds to the intensity of each sensation. Both threshold and intensity will be measured in the peroneal nerve territory in all subjects, and at one other variable place, which will be matched 1:1 between patients and controls. The variable spot will consist of a patient's sensory tic site. Next, EMG activity will be measured from up to 8 muscles in the area of a sensory tic. Patients will report when a sensory tic is occurring, and will be asked to resist the motor tic for at least 12 seconds from that point. Total EMG activity will be measured in muscles surrounding the sensation at 1, 4, and 7 seconds before and after the tic.

OUTCOME MEASURES:

Outcome measures include the sensory threshold values for olfaction and touch and the reported intensity values. The outcome measures of the EMG study include the power of total EMG activity at time points before and after a tic.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers ages 18 to 65 who have who have given their consent.

Patients will be ages 18 to 65 and have clinically documented Tourette's syndrome or chronic motor tic disorder as defined by DSM-IV-TR (American Psychiatric Association, 2000) and evaluation of tic severity using the Yale Tic Scale (YGTS). This criterion will be established by preliminary screening in the NINDS Movement Disorders Outpatient Clinic. Structure Clinical Interview for (DSMIV SCID) will be administered to all patients to ensure that strict DSM-IV criteria for Tourette Syndrome have been met and to assess for possible comorbid psychiatric disorders.

Patients with at least moderate premonitory urge, as evaluated with the PUTS.

EXCLUSION CRITERIA:

Subjects younger than 18 or older than 65 years.

Subjects with 1) major depression, 2) bipolar disorder, or 3) psychotic disorder.

Subjects who are unable to abstain from alcohol or any psychiatric medications 24 hours prior to the study.

Subjects with acute or chronic upper respiratory illness, nasal allergies, or subjects using medications to treat these conditions, including antihistamines, nasal topical steroids, vasoconstrictor nasal sprays, or normal saline sprays.

Women who are pregnant.

Individuals with Restless Legs syndrome.

Individuals with a diagnosis of peripheral neuropathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-08-21; Study Completion 2011-05-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bartoshuk LM, Duffy VB, Green BG, Hoffman HJ, Ko CW, Lucchina LA, Marks LE, Snyder DJ, Weiffenbach JM. Valid across-group comparisons with labeled scales: the gLMS versus magnitude matching. Physiol Behav. 2004 Aug;82(1):109-14. doi: 10.1016/j.physbeh.2004.02.033. PMID 15234598
- [Background] Bliss J. Sensory experiences of Gilles de la Tourette syndrome. Arch Gen Psychiatry. 1980 Dec;37(12):1343-7. doi: 10.1001/archpsyc.1980.01780250029002. PMID 6934713
- [Background] Garcia-Perez MA. Forced-choice staircases with fixed step sizes: asymptotic and small-sample properties. Vision Res. 1998 Jun;38(12):1861-81. doi: 10.1016/s0042-6989(97)00340-4. PMID 9797963